CLINICAL TRIAL: NCT02718586
Title: Association of Serum Myokines and Protein Energy Wasting, Inflammation and Atherosclerotic Vascular Disease in Hemodialysis Patients
Brief Title: Serum Level of Myokines and Protein Energy Wasting, Inflammation and Atherosclerosis in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Principal Investigator, Paik Seong Lim, Director, Tungs' Taichung Metroharbour Hospital
Other Study IDs: 104074
Record Dates: First submitted 2016-03-04; First posted 2016-03-24 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Protein-energy; Imbalance
Keywords: Myokines; Protein Energy Wasting; Hemodialysis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim is to test if serum level of myokines are associated with protein energy wasting, inflammation and atherosclerotic vascular disease among Taiwanese dialysis patients. Some novel myokines levels, anthropometric parameters, cardiovascular risk factors, and presence of endothelial dysfunction will be examined in 250 subjects. The distribution of some recently identified myokines such as irisin, myotatin etc levels will be studied and correlated markers of malnutrition, endothelial dysfunction, inflammation and insulin resistance. In the present study, the investigators will further follow and investigate whether serum myokines levels are associated with long-term mortality from all causes and from cardiovascular disease.

DETAILED DESCRIPTION:
Study Design and Population

In this study, patients who underwent stable hemodialysis at least 3 months at Tung Taichung Metroharbor Hospital will be enrolled. Baseline clinical data such as age, sex, height, bodyweight , clinical etiology of Chronic kidney disease(CKD) if possible, comorbidities, blood pressure, laboratory measures [such as serum creatinine, albumin, C-reactive protein (CRP), total cholesterol, complete blood counts, urine routines, anthropometric information and various potential indicators of protein energy wasting [such as body mass index, waist/hip ratio, mid-arm circumference (MAC), triceps skinfold thickness (TSF), mid-arm muscle circumference (MAMC), mid-arm muscle area (MAMA), SGA, BIS analyses, dual energy x-ray absorptiometry(DEXA),handgrip (HG)] will be collected. For the laboratory tests, fasting blood and urine samples are obtained from each patient and performed by means of routine methods in the investigators hospital. All patients received echocardiograms studies performed within 3 months after enrollment, which were used to estimate congestive heart failure(CHF, defined as an ejection fraction of <50%) or left ventricular hypertrophy (LVH, defined as left ventricle mass index >125 g/m2 in men and 100 g/m2 in women).Cardiovascular disease( CVD) was defined as a previous history of CHF, LVH, ischemic heart disease(including prior history of angina, myocardial infarction, coronary artery bypass grafting and percutaneous cardiac catheter intervention) or cerebrovascular disease (including prior history of transient ischemic attack and stroke). Information about conventional clinical risk factors, such as smoking, diabetes mellitus, hypertension, medication and other necessary data at baseline will be obtained from a standardized interview and examination. The diagnosis of type 2 diabetes is made according to the criteria of the American Diabetes Association.

Patients with malignant disease, acute infectious disease, inflammatory disease (such as collagen disease), advanced liver disease, and those taking any type of immunosuppressive medication were also excluded. Patients with clinical manifestations of atherosclerosis, congestive heart failure, history of stroke, a previous history of coronary intervention or coronary artery bypass graft surgery, and presence peripheral vascular disease were recorded.

Anthropometrics, and Handgrip Strength

Body weight was measured with light clothing on up to 0.1 kg. Height was measured up to 0.1 cm. Waist circumference was measured at the midpoint between upper iliac and lower costal level up to 0.1 cm at the end of normal expiration. Hip circumference was measured around the largest part of the hip. Anthropometric measurements were obtained immediately after the HD session by a trained researcher. Body mass index (BMI) was calculated as body mass divided by stature squared. The International Society of Renal Nutrition and Metabolism(ISRNM) panel recommends that a BMI lower than 23 kg/m2 is a marker of Protein Energy Wasting(PEW). Anthropometric measurements include TSF used skinfold calipers; MAC measured by a stretchable measuring tape, MAMC equals MAC(centimeter) - 3.14 x TSF (millimeter)/10 and MAMA equals (MAMC2/4π). Muscle mass area (MMA) was calculated using the following equation: MMA = ([MAC {cm} - π x triceps skinfold {cm}]2/4π) -n, where n = 10 for men and 6.5 for women . Muscle strength as hand grip strength (HGS) test was measured by Hand Dynamometer. HGS was measured 3 times for both left and right hands with patients in a standing position using a dynamometer in units of kilograms. Patients held the dynamometer at thigh level and were encouraged to squeeze the instrument as hard as possible for 3 s. The maximum grip strength among all measurements was used for this study. Three sets of measurements at each site were averaged and used in the analyses.

Malnutrition Inflammation Score

To assess the malnutrition-inflammation complex syndrome(MICS), also known as the Kalantar score, developed, and validated by Kalantar- Zadeh et al. was measured at baseline. The Malnutrition-Inflammation Score(MIS) has ten components [change in end dialysis dry weight, dietary intake, gastrointestinal symptoms, functional capacity, comorbidities, decreased fat stores or loss of subcutaneous fat (according to SGA), signs of muscle wasting (according to SGA), BMI, serum albumin, and total iron binding capacity], each with four levels of severity, from 0 (normal) to 3 (severely abnormal). The sum of the MIS components ranges from 0 (normal) to 30 (severely malnourished), in which a higher score reflects greater malnutrition and inflammation severity.

The comorbidity component was scored as 0 if no comorbidities were present; 1 if there were mild comorbidities present and major comorbid conditions (MCCs) were absent (such as New York Heart Association Class III or IV congestive heart failure, severe coronary artery disease, acquired immunodeficiency syndrome, moderate- to-severe chronic obstructive pulmonary disease, and metastatic malignancies); 2 if moderate comorbidities were present, including one MCC; and 3 if multiple severe comorbidities were present, including two or more MCCs. Subjective global assessments (SGAs) were performed by an experienced physician according to conventional SGA guidelines.

Dual-energy X-ray absorptiometry

Whole-body scans are performed according to manufacturer's instructions, and body fat, lean tissue mass (LTM) and bone mineral content (BMC) are analysed using the manufacturer's software. DEXA estimate of fat-free mass (FFM) was calculated as a sum of LTM and BMC estimates. All patients were examined by the same observer.

Bioelectric impedance spectroscopy (BIS)

BIS measurement was performed in each of the participants enrolled in the study by a specific member of staff who had completed a training course in the BIS technique, using a portable whole body bioimpedance spectroscopy device, the body composition monitor. The body composition monitor(BCM) measures the impedance spectroscopy at 50 different frequencies between 5 kilohertz(kHz) and 1 megahertz (MHz). Measurements were taken on the midweek dialysis session before the start of the hemodialysis treatment with the patient calm, supine, and relaxed in the dialysis bed for 10 minutes. Specific exclusion criteria were dictated by the device and included history of a pacemaker, defibrillator, metallic sutures, or stent implantation and amputation of a major limb.

Biochemical Analysis

Blood samples were taken in a nonfasting state before a midweek hemodialysis session. Complete blood count, creatinine, urea, albumin, transferrin, total carbon dioxide, hsCRP , triglycerides (TG), total cholesterol (TC), high-density lipoprotein-cholesterol (HDL-C), low-density lipoprotein-cholesterol (LDL-C), and fasting blood glucose are measured by routine laboratory methods. Another blood samples will be stored at -80 degree centigrade for subsequent assay of items such as insulin, interleukin-6, pentraxin, nitrotyrosine for markers of endothelial dysfunction such as Asymmetric dimethylarginine( ADMA), adropin and insulin resistance (adiponectin, resistin and leptin). Homeostatic Model Assessment Insulin Resistance(HOMA-IR) was calculated as fasting insulin (U/l) × fasting glucose (mg/dl)/405, as described by Matthews et al.

Serum total p-cresol and indoxyl sulfate (i.e. combined free and protein-bound fractions) were analyzed with High-performance liquid chromatography (HPLC). Briefly, serum samples were deproteinized for the determination of indoxyl sulfate by the addition of three parts methanol to one part serum. Total p-cresol (i.e. the combined free and protein-bound fraction) was analysed after deproteinization (acid and heat) and extraction (ethyl acetate) of serum samples.

Measurement of serum myostatin, irisin and myonectin

Serum myostatin levels are measured with a competitive immunoassay kits according to the manufacturer's protocol. Serum irisin concentration was measured using the enzymelinked immunosorbent assay). The assay was proven to be highly sensitive to human irisin. Serum myonectin (Circulating Complement-C1q Tumor necrosis factor(TNF)-Related Protein 15) Serum myonectin was determined with a commercially available enzyme-linked immunosorbent assay kit.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged between 20-70 years.
* Received stable hemodialysis at least 3 months.
* Written informed consent.

Exclusion Criteria:

* Patients with malignant disease, acute infectious disease, inflammatory disease (such as collagen disease), advanced liver disease, and those taking any type of immunosuppressive medication are excluded.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis (HD) patients
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Presence of protein energy wasting | 1 year
  According to the diagnostic criteria for PEW proposed by ISRNM

IPD SHARING:
Plan to Share IPD: Yes